CLINICAL TRIAL: NCT06912997
Title: Effects of Inspiratory Muscle Training on Hemodynamic and Cerebrovascular Responses During Maintenance of Postural Balance in Parkinson's Disease
Brief Title: Effects of Inspiratory Muscle Training on Parkinson's Disease
Acronym: IMT_PD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Gabriel Dias Rodrigues, PhD and Visiting Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 58755522.5.0000.5243
Record Dates: First submitted 2025-03-19; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Neurodegenerative disease; Movement disorder; Postural balance; respiratory training; inspiratory training; Physical exercise; Cerebrovascular control; blood pressure; cardiovascular autonomic control
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Movement Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A training group and a placebo group (sham)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The home-based inspiratory muscle training (IMT) protocol in experimental group will use an inspiratory threshold loading device (PowerBreathe Wellness, Southam, United Kingdom). IMT for experimental group will start with a minimal load (~9 cmH2O) during the first week, aiming for a familiarization process. During the second week, the IMT targeted a moderate load of 45% of maximal inspiratory pressure (MIP) previously defined, which will be gradually increased by 10% of MIP each week until reaching 75% of MIP in the final week.
  Interventions: Other: Exercise
- Sham group (Sham Comparator): The Sham group will performer the same training protocol that experimental group, but at 5% of MIP during all weeks. Therefore, the sham group will not increase the training load during the protocol.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Other: Exercise — The home-based inspiratory muscle training (IMT) protocol will use an inspiratory threshold loading device (PowerBreathe Wellness, Southam, United Kingdom). IMT for experimental group will start with a minimal load (~9 cmH2O) during the first week, aiming for a familiarization process. During the second week, the IMT targeted a moderate load of 45% of maximal inspiratory pressure (MIP) previously defined, which will be gradually increased by 10% of MIP each week until reaching 75% of MIP in the final week.
  Arms: Experimental group
Other: Sham Comparator — The Sham group will performer the same training protocol that experimental group, but at 5% of MIP during all weeks. Therefore, the sham group will not increase the training load during the protocol.
  Arms: Sham group

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative movement disorder that provoke motors and non-motors symptoms causing further dependence and disability. Among non-motor issues, orthostatic hypotension (OH) is a severe manifestation of autonomic dysfunctions, occurring in approximately 30% of those with PD. The fall in blood pressure (BP) during orthostatic position (ORT) is normally compensated to maintain adequate cerebral blood flow (CBF) through autoregulation of cerebral vessels (AC). However, if AC is compromised, CBF may decrease and cause pre-syncope symptoms such as dizziness and loss of balance. Inspiratory muscle training (IMT) is a non-pharmacological strategy to improve respiratory muscle strength, cerebrovascular, cardiovascular control in several populations. However, the effects of IMT on cardiovascular autonomic control (i.e. baroreflex sensitivity-BRS), hemodynamic and AC during ORT in PD patients with and without orthostatic hypotension have not yet been studied. Our hypothesis is that IMT will increase inspiratory muscle strength and influence spontaneous breathing pattern, improving BRS. In addition, IMT will cause a smaller drop in BP and CBF during ORT. Furthermore, maintaining CBF will reduce postural instability during ORT. PD patients without and with OH (PD-OH) will participate in the study and will be randomly divided into two groups recruited at the Antônio Pedro University Hospital. The experimental group will perform 6-8 weeks of training at 30-75% of maximum inspiratory pressure (MIP), and the placebo group will perform the same training protocol at 5% of MIP (sham). The home-based protocol will be of 30 repetitions twice a day, five days a week. In active ORT test, BP, R-R intervals, stroke volume, cardiac output, respiratory rate, ventilatory variables and mean cerebral blood flow velocity (MCAv) will be continuously monitored for 10 minutes in the supine position (SUP), 10 minutes in the sitting position and then 6 minutes in the ORT position. Oscillations of the body's center of pressure (COP), through a force platform, and neuromuscular responses of the gastrocnemius and tibialis anterior muscles, through surface electromyography, will be recorded while maintaining the ORT position. The orthostatic test will be performed before and after the interventions (placebo and experimental). We believe that IMT will promote an improvement in BRS, AC, and postural control, presenting itself as a potential non-pharmacological countermeasure in autonomic dysfunctions and in the prevention of falls in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD according to Movement Disorder Society (MDS) criteria
* treatment at Antonio Pedro Hospital (HUAP) for >6 months;
* stable Parkinson's medication for at least 30 days prior to testing.

Exclusion Criteria:

* active smokers or those who quit <5 years ago
* pulmonary or cardiovascular complications in the past 3 months
* arrhythmias or beta-blocker use
* Both groups required spirometry values >80% of predicted age

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
center of pressure of the body | Two measurements will be taken: one at baseline (second visit) and after 6 weeks of training (third visit)
  The variables related to postural balance will be performed on a force platform (Accusway Dual Top, USA) in a bipedal position. The participants' feet will be positioned with the heels together and with a 30° gap between the feet. Throughout the test, the individual's center of pressure (COP) will be continuously recorded, determined as a neuromuscular response to the location of the center of gravity (COG). The starting point used for the assessment will be considered the moment when the individual reaches the orthostatic position, for which the highest value of the weight force (Fz) will be obtained. The elliptical area, the total distance and the displacement speed COPxy will be calculated as COP variables. The signals will be filtered at a frequency of 50 Hz as a Hamming window and a "low-pass" filter to reduce interference.

SECONDARY OUTCOMES:
cerebral blood flow | Two measurements will be taken: one at baseline (second visit) and after 6 weeks of training (third visit)
  In order to estimate changes in cerebral perfusion, the blood flow velocity in the middle cerebral artery (MCAv) will be used, insonated using a pulsed transcranial ultrasound Doppler with 2-MHz waves. The transducer will be positioned over the right temporal window in all participants, fixed with an adjustable headband. The insonation depth will be 20 and 60 mm, depending on the anatomical positioning of the vessel, to ensure the best signal quality. The cerebral vascular conductance index (CVCi) will be calculated as the mean of the MCAv divided by the mean arterial pressure (MAP) obtained through photoplethysmography. This index will be used as a way to estimate changes in cerebrovascular conductance.Cerebral autoregulation will be dynamically assessed by the cerebral autoregulation index (RoR), calculated using the following formula: RoR = (ΔCVCi/ΔT)/ΔMAP. The first field of the formula consists of a linear regression between CVCi and time. The delta MAP will be obtained.
Hemodynamic variables | Two measurements will be taken: one at baseline (second visit) and after 6 weeks of training (third visit)
  Blood pressure will be recorded beat-to-beat using infrared photoplethysmography (FinometerPro; Finapres Medical Systems, Arnhem, The Netherlands), R-R intervals using electrocardiography (Equivital, ADinstruments, AUS), and stroke volume and cardiac output will be recorded noninvasively using transthoracic impedance (PhysioFlow, PF-05, Manatec Biomedical, Macheren, France). All variables will be recorded simultaneously at a sampling rate of 1 kHz and analyzed offline using a data acquisition system and data analysis software (PowerLab 16SP hardware and LabChart 8 PRO software; ADInstruments, Australia).
Metabolic and Ventilatory Variables | Two measurements will be taken: one at baseline (second visit) and after 6 weeks of training (third visit)
  Metabolic and ventilatory variables will be acquired by a metabolic gas analyzer (Ultima CPX; Medgraphics, St. Paul, MN, USA) and a medium-flow pneumotachograph (Medgraphics, St. Paul, MN, USA). The device will be calibrated at the beginning of each test using a 3-L cylinder. The variables recorded will be minute ventilation (VE), tidal volume (Vt), expired carbon dioxide pressure (PetCO2), expiratory time (Te), inspiratory time (Ti), the ratio between Ti and total respiratory time (Ti/Ttot) and between Vt and Ti (Vt/Ti).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal Fluminense, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No